CLINICAL TRIAL: NCT04873349
Title: Assessment of the Clinical Effectiveness of Standardized Olive Leaf Capsules; as a Co-therapy in the Treatment of Non-hospitalized COVID-19 Patients; a Randomized Clinical Trial
Brief Title: Standardized Olive Leaf Capsules; as a Co-therapy in the Treatment of COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shimaa M. Abdelgawad (Other)
Responsible Party: Sponsor-Investigator, Shimaa M. Abdelgawad, Assisting lecturer, Pharmacognosy Department, Faculty of Pharmacy, Fayoum University, Egypt, Fayoum University
Organization: Fayoum University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 2121
Record Dates: First submitted 2021-05-04; First posted 2021-05-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Covid19; COVID-19 Respiratory Infection; Symptoms and Signs; COVID-19 Acute Bronchitis; Disseminated Intravascular Coagulation
Keywords: COVID-19, Infection, Bronchitis, Coagulation, Symptoms
MeSH Terms: conditions — COVID-19; Signs and Symptoms; Disseminated Intravascular Coagulation; Infections; Bronchitis; Thrombosis | interventions — oleuropein

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Olive leaf capsules (Active Comparator): Non-hospitalized COVID-19 patients who have positive PCR results and show mild to moderate clinical manifestations and symptoms (20-30 patients) will receive a 50% standardized olive leaf capsule 750 mg (700 mg oleuropein/day; the active principle in olive leaf) two times daily for a period of ten days alongside with the Egyptian protocol medications. All the active comparator participants should be adults, with no chronic diseases (except hypertension and diabetes), non addict or alcoholics.
  Interventions: Dietary Supplement: Nusapure standardized olive leaves capsule, 750 mg (50% oleuropein)
- Starch capsules (Placebo Comparator): Non-hospitalized COVID-19 patients who have positive PCR results and show mild to moderate clinical manifestations and symptoms (20-30 patients) will receive a placebo starch capsules (750 mg) two times daily for a period of ten days alongside with the Egyptian protocol medications. All the placebo comparator participants should be adults, with no chronic diseases (except hypertension and diabetes), non addict or alcoholics.
  Interventions: Dietary Supplement: Nusapure standardized olive leaves capsule, 750 mg (50% oleuropein)

INTERVENTIONS:
Dietary Supplement: Nusapure standardized olive leaves capsule, 750 mg (50% oleuropein) — two study groups; test group will receive Nusapure standardized olive leaves capsule, 750 mg (50% oleuropein) while placebo group will receive starch group

SUMMARY:
Starting from December 2019, novel coronavirus disease 2019 (COVID-19) pandemic has caused a tremendous economic loss and unprecedented health crisis across the globe. Discovering an effective and safe drug candidates for the treatment of COVID-19 and its associated symptoms became a global urgent demand especially due to limited data that have been released regarding the vaccine efficacy and safety in humans. Reviewing the recent research, Olive leaf was selected as a potential co-therapy supplement for the treatment and the improvement of clinical manifestations in COVID-19 patients. Olive leaves reported to be rich in phenolic compounds such as oleuropein, hydroxy tyrosol, verbascoside, apigenin-7-glucoside and luteolin-7-glucoside which has been reported as anti-SARS-CoV-2 metabolites in recent In silico, computational and in vitro studies. In addition, olive leaf extract was previously reported in several in vivo studies for its anti-inflammatory, analgesic, antipyretic, immunomodulatory and anti-thrombotic activities which is of a great benefit in the control of associated inflammatory cytokine storm and disseminated intravascular coagulation in COVID-19 patients.

A placebo-controlled, randomized clinical trial at Fayoum University Hospital in Egypt will be conducted. RT-PCR confirmed COVID-19 adults showing mild to moderate disease will be enrolled in the study. Patients presenting with multi-organ failure, ventilator support, and chronic diseases (except diabetes mellitus and hypertension) were excluded. Patients were randomly assigned in 1:1 ratio to receive standardized olive leaves capsules (containing 20-50% oleuropein) or placebo up-to 10 days along with standard care. The expected outcomes included symptom alleviation, viral clearance, improvement of analysis (CBC, CRP, LDH, ESR, Ferritin, D-dimer, creatinine, ALT and AST) and a 10-day mortality in intention-to-treat population.

DETAILED DESCRIPTION:
Objectives:

We will evaluate the efficacy of standardized olive leaf capsules as additive therapy to the standard therapeutic regimen (for a period 10 days) on clinical symptoms, viral clearance, improvement of analysis:

1. Complete blood count (CBC).
2. C-Reactive Protein (CRP)
3. Lactate dehydrogenase (LDH).
4. Erythrocyte Sedimentation rate (ESR).
5. Serum Ferritin
6. D-dimer
7. Serum creatinine.
8. Alanine Amino Transferase (ALT) and Aspartate Amino Transferase (AST).
9. Also, a 30-day mortality in patients with confirmed COVID-19, who are mild to moderately ill.

Trial design:

This is a single-center, randomized, double-blind, placebo-controlled clinical trial with a parallel-group design conducted at Fayoum university Hospital, Fayoum, Egypt.

Research Plan and Methodology 1-Complete patient history will be recorded (other diseases, current medications, age, sex, etc.) 2-Clinical investigation of patients by the physicians at Chest Department, Fayoum University Hospital including measurements such as Temperature and Oxygen saturation.

3-Patients will be tested for infection by PCR and all patients to be enrolled at the study should show positive PCR result.

4-The following analysis will be carried out for all the patients included in the study; CBC, CRP, LDH, ESR, Ferritin, D-dimer, creatinine, ALT and AST before treatment and for follow up after 10 days.

Participants:

All outpatients admitted to Chest Diseases Departments of Fayoum university Hospital, will be screened for the following criteria.

Inclusion criteria:

1. Adults.
2. Confirmed SARS-CoV-2 diagnosis (positive polymerase chain reaction by nasopharyngeal swab).
3. Mild to Moderate COVID-19 patients.
4. No history of the current use of olive leaf capsules supplement.

Exclusion criteria:

1. Severe and critical COVID-19 patients who need hospitalization.
2. Patients need ventilatory support or showing chronic obstructive pulmonary disease (COPD).
3. Patients showing any chronic disease (except hypertension and diabetes mellitus).
4. Patients who have multiorgan failure.

3. Use of alcohol, other investigational medicines, and illegal drugs (during the last 30 days).

Intervention and comparator:

A total of 60 patients randomized into two groups (30 in each group). The patients will be divided into 2 groups Intervention group: All patients receive the standard treatment regimen for COVID-19, according to the Egyptian Ministry of Health protocol, along with 2-3 capsules/day of standardized olive leaf containing 20-50% oleuropein (500-750 mg oleuropein daily) for a period of ten days.

Control group: The standard therapeutic regimen for COVID-19 along with placebo capsules daily for a period of ten days.

Main outcomes:

The main outcomes are the improvement of clinical symptoms, as well as oxygen saturation, viral clearance, improvement of analysis (CBC, CRP, LDH, ESR, Ferritin, D-dimer, creatinine, ALT and AST) within 10 days of randomization in patients with confirmed COVID-19, who are mild to moderately ill.

Randomization:

Included patients will be allocated to one of the study arms using block randomization in a 1:1 ratio (each block consists of 10 patients). This randomization method ensures a balanced allocation between the arms during the study. A web-based system will generate random numbers for the allocation sequence and concealment of participants. Each number relates to one of the study arms.

Ethical considerations All participants should Sign informed consent and show willingness to accept randomization to any assigned treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Adults.
2. Confirmed SARS-CoV-2 diagnosis (positive polymerase chain reaction by nasopharyngeal swab).
3. Mild to Moderate COVID-19 patients.
4. No history of the current use of olive leaf capsules supplement.

Exclusion Criteria:

1. Severe and critical COVID-19 patients who need hospitalization.
2. Patients need ventilatory support or showing chronic obstructive pulmonary disease (COPD).
3. Patients showing any chronic disease (except hypertension and diabetes mellitus).
4. Patients who have multiorgan failure.

3. Use of alcohol, other investigational medicines, and illegal drugs (during the last 30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Improving the clinical symptoms in mild to moderate COVID -19 patients | 10 days after treatment
  It is expected that the examined drug will alleviate symptoms such as fever, cough, sore throat and muscles ache
Viral clearance in mild to moderate COVID -19 patients | 10 days after treatment
  It is expected that the examined drug will make the Polymerase chain reaction (PCR ) results for the test group negative within 10 days of treatment
Improvement of analysis (CBC) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group such as increase lymphocyte count in complete blood count (CBC).
Improvement of analysis (CRP) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of C-reactive protein (CRP).
Improvement of analysis (LDH) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of Lactate dehydrogenase (LDH).
Improvement of analysis (ESR) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of Erythrocyte sedimentation rate (ESR).
Improvement of analysis (Ferritin) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of Ferritin.
Improvement of analysis (D-dimer) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of D-dimer.

SECONDARY OUTCOMES:
Evaluate mortality rate in patients with confirmed COVID-19 moderately ill | 10 days after treatment
  It is expected that the drug will reduce the conversion in cases from moderate to sever cases and so decrease the mortality rate
Improvement of analysis (creatinine) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of creatinine.
Improvement of analysis (ALT) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of Alanine Amino Transferase (ALT).
improvement of analysis (AST) | 10 days after treatment
  It is expected that the treatment will improve the lab analysis for treatment group and prevent elevation and/or decrease the elevated values of Aspartate Amino Transferase (AST).

CONTACTS AND LOCATIONS:
Locations (1):
- Shimaa Abdelgawad, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No